CLINICAL TRIAL: NCT01073462
Title: Postmarketing Observational Study to Evaluate the Effect of Zemplar (Paricalcitol IV) on Cardiac Morbidity in Patients With Chronic Kidney Disease Stage 5 Over 2 Years.
Brief Title: Study to Evaluate the Effect of Intravenous (IV) Paricalcitol (Zemplar) on Cardiac Morbidity in Patients With Chronic Kidney Disease (CKD) Stage 5 Over 2 Years
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Assign Data Management and Biostatistics GmbH (Other)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-680
Record Dates: First submitted 2010-02-20; First posted 2010-02-23 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease Stage V; Cardiac Morbidity
Keywords: Secondary Hyperparathyroidism (sHPT); Paricalcitol; Chronic kidney disease stage 5 (CKD stage 5)
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Paricalcitol IV: Participants with chronic kidney disease stage 5 with secondary hyperparathyroidism and cardiac morbidity received intravenous (IV) paricalcitol (Zemplar) prescribed according to current practice with regards to dose, population and indication for up to 2 years.

SUMMARY:
The purpose of this study was to ascertain the percentage of cardiac patients with chronic kidney disease (CKD) stage 5 treated with paricalcitol IV achieving intact parathyroid hormone (iPTH) levels in target range of Kidney Disease Outcomes Quality Initiative (K/DOQI) treatment guidelines (150 - 300 pg/mL) after 2 years.

DETAILED DESCRIPTION:
Secondary hyperparathyroidism (SHPT) is a frequent complication in patients with chronic kidney disease (CKD) stage 5 receiving dialysis. SHPT is an adaptive response to CKD and is characterized by an elevation in parathyroid hormone (PTH) and consecutively high calcium levels. Elevations in calcium levels, phosphate levels, and PTH are correlated with CKD disease progression as well as development or aggravation of cardiovascular impairment. Many CKD patients cannot be treated well with Vitamin D analogues because of effects on calcium. Hypercalcemia is a well - known factor for cardiac disease. No data are available in Austria for a cohort with cardiac disease treated with Zemplar (paricalcitol IV).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years
* Patients with secondary hyperparathyroidism associated with CKD stage 5, serum iPTH > 150 pg/mL,
* Cardiac disease as described by Medical Dictionary for Regulatory Activities (MedDRA) terms:

  * cardiac disorder as cardiac arrhythmias
  * cardiac disorder signs and symptoms
  * cardiac neoplasm
  * cardiac valve disorder
  * heart failures
  * myocardial disorder
  * pericardial disorder
  * Serum phosphate level < 6.5 mg/dL and serum calcium level < 10.5 mg/dL

Exclusion Criteria:

* Patients who meet contraindications as outlined in the latest version of Zemplar (Paricalcitol IV) summary of product characteristics
* Patients with known hypersensitivity to paricalcitol or any component of the formulation, vitamin D intoxication, hypercalcemia; cinacalcet as concomitant medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigational sites were clinic centers with experience in the treatment of chronic kidney disease stage 5 patients and hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Dworan-Timler, Study Director — AbbVie Austria
Locations (12):
- Austria (12):
  - Site Reference ID/Investigator# 27447, Graz
  - Site Reference ID/Investigator# 49182, Graz
  - Site Reference ID/Investigator# 27483, Graz
  - Site Reference ID/Investigator# 52742, Graz
  - Site Reference ID/Investigator# 27487, Innsbruck
  - Site Reference ID/Investigator# 36983, Linz
  - Site Reference ID/Investigator# 27484, Linz
  - Site Reference ID/Investigator# 27485, Rottenmann
  - Site Reference ID/Investigator# 27446, Vienna
  - Site Reference ID/Investigator# 53469, Vienna
  - Site Reference ID/Investigator# 27482, Vienna
  - Site Reference ID/Investigator# 10981, Vienna

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paricalcitol IV
Started | 67
Completed | 26
Not Completed | 41
Not completed — Death | 14
Not completed — Kidney transplant | 10
Not completed — Low parathyroid hormone levels | 8
Not completed — Serious adverse event | 2
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 40
Region of Enrollment [Number; unit: participants]
  Austria | 67
Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Blood pressure data were available for 66 participants
  mm Hg
    Systolic | 137.2 (19.4)
    Diastolic | 75.1 (11.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Intact Parathyroid Hormone (iPTH) Level Within the Target Range
Description: Target range of intact parathyroid hormone was defined according to the Kidney Disease Outcomes Quality Initiative (K/DOQI) treatment guidelines as between 15.9 - 31.8 pmol/L (150 to 300 pg/mL).
Time Frame: Baseline and Months 3, 6, 12, 18, and 24
Population: Intent-to-treat population; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
percentage of participants
  Baseline | 28.4
  Month 3 | 43.3
  Month 6 | 35.8
  Month 12 | 38.8
  Month 18 | 37.3
  Month 24 | 35.8

2. Secondary Outcome: Percentage of Participants With Hypercalcemia
Description: Hypercalcemia was defined as a calcium value of > 2.625 mmol/L (10.5 mg/dL) in one measurement. Serum calcium was measured at every study visit.
Time Frame: Baseline and Months 3, 6, 12, 18, and 24
Population: Intent-to-treat; LOCF was used
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
percentage of participants
  Baseline | 0.0
  Month 3 | 0.0
  Month 6 | 0.0
  Month 12 | 1.5
  Month 18 | 0.0
  Month 24 | 1.5

3. Secondary Outcome: Percentage of Participants With Hyperphosphatemia
Description: Hyperphosphatemia was defined as a phosphate value of > 2.1 mmol/L (6.5 mg/dL) in one measurement. Serum phosphate was measured at every study visit.
Time Frame: Baseline and Months 3, 6, 12, 18, and 24
Population: Intent-to-treat; LOCF was used. "n" indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
percentage of participants
  Baseline (n=65) | 0.0
  Month 3 (n=67) | 28.4
  Month 6 (n=67) | 31.3
  Month 12 (n=67) | 25.4
  Month 18 (n=67) | 23.9
  Month 24 (n=67) | 22.4

4. Secondary Outcome: Percentage of Participants With at Least a 30%-Reduction in iPTH Levels
Description: The percentage of participants with at least a 30% reduction in intact parathyroid hormone (iPTH) levels from Baseline level.
Time Frame: Baseline and Months 3, 6, 12, 18, and 24
Population: Intent-to-treat; LOCF was used.
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
percentage of participants
  Month 3 | 41.8
  Month 6 | 40.3
  Month 12 | 47.8
  Month 18 | 52.2
  Month 24 | 47.8

5. Secondary Outcome: Percentage of Participants With at Least 30%-Reduction in iPTH Levels in at Least Two Consecutive Measurements
Description: The percentage of participants with at least a 30% reduction in intact parathyroid hormone (iPTH) level from Baseline in at least 2 consecutive visits.
Time Frame: Baseline to Month 24
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
percentage of participants | 44.8

6. Secondary Outcome: Percentage of Participants With at Least One Concomitant Medication
Description: The percentage of participants with at least one concomitant medication during the course of the study, by the following types:
  * Phosphate binder
  * Epoetin
  * Renin-Angiotensin-Aldosterone System (RAAS) inhibitors
  * Cinacalcet
  * Other
Time Frame: 24 months
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
percentage of participants
  Phosphate binder | 80.6
  Epoetin | 68.7
  RAAS Inhibitor | 43.3
  Cinacalcet | 13.4
  Other | 86.6

7. Secondary Outcome: Percentage of Participants Experiencing Hospitalization
Description: The percentage of participants with at least one hospitalization, at least one cardiac-related hospitalization and at least one non-cardiac-related hospitalization during the course of the study.
Time Frame: 24 months
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
percentage of participants
  Hospitalizations | 41.8
  Cardiac-related hospitalizations | 14.9
  Non-cardiac-related hospitalizations | 37.3

8. Secondary Outcome: Number of Participants With Cardiac Disease Progression
Description: Cardiac disease progression was determined by the Investigator.
Time Frame: Month 3, 6, 12, 18, and 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Paricalcitol IV
Number analyzed (Participants) | 67
participants
  Month 3 | 2
  Month 6 | 2
  Month 12 | 4
  Month 18 | 0
  Month 24 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Paricalcitol IV
Serious Adverse Events (participants affected / at risk) | 31/67
Other Adverse Events (participants affected / at risk) | 23/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol IV (N=67)
Cardiac failure (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 3
Acute tonsillitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Muscle abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pancreatic abscess (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 5
Multiple fractures (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Carotid artery stenosis (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Death (General disorders) | 3
Knee arthroplasty (Surgical and medical procedures) | 1
Medical device implantation (Surgical and medical procedures) | 1
Stent placement (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Vertigo (Ear and labyrinth disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol IV (N=67)
Hyperphosphataemia (Metabolism and nutrition disorders) | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Cardiac valve disease (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.